CLINICAL TRIAL: NCT01121055
Title: Effect of Additive Lorazepam on Patient Satisfaction as a Premedication in Diagnostic Flexible Bronchoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seok-Chul Yang, MD, PhD, FCCP, Division of Pulmonology and Critical Care Medicine, Department of Internal Medicine and Lung Institute of Medical Research Center, Seoul National University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Lorazepam in FB
Record Dates: First submitted 2010-05-09; First posted 2010-05-12 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Patient Satisfaction for Bronchoscopy
Keywords: Fiberoptic Bronchoscopy; Patient; Satisfaction; Lorazepam
MeSH Terms: conditions — Personal Satisfaction | interventions — Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Placebo 1T by mouth (po) at night one day before FB and placebo 1T po 30min before the FB
  Interventions: Drug: Control
- Lorazepam (Experimental): Lorazepam 0.5mg po at night one day before FB and Lorazepam 1mg po 30min before the FB
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Lorazepam — Lorazepam 0.5mg po at night one day before FB and Lorazepam 1mg po 30min before the FB
  Arms: Lorazepam
Drug: Control — Placebo 1T po at night one day before FB and placebo 1T po 30min before the FB
  Arms: Control

SUMMARY:
Many patients undergoing flexible bronchoscopy (FB) experience anxiety and discomfort during the procedure. The investigators want to evaluate whether an additional Lorazepam premedication would improve patient satisfaction for FB.

DETAILED DESCRIPTION:
The enrolled patients are randomized to either the control or Lorazepam groups according to a random sample chart of numbers. The patients complete questionnaires about baseline anxiety level and satisfaction for FB within 24 hours after the FB.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years or older) admitted to the Respiratory Department

Exclusion Criteria:

* outpatient procedures
* therapeutic bronchoscopy
* expected operation or discharge within 24 hours after the FB
* sedative premedication
* endotracheal intubation with mechanical ventilation
* inability to speak Korean

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-08 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | within 24 hr of bronchoscopy

SECONDARY OUTCOMES:
relationship between patient satisfaction and sleep quality, anxiety level | 24hr before and after bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Chul Yang, MD, Study Chair — Division of Pulmonology and Critical Care Medicine, Department of Internal Medicine and Lung Institute of Medical Research Center, Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea